CLINICAL TRIAL: NCT07098923
Title: The Effect of Combined Aerobic and Resistance Exercise on Blood Pressure Variability on Peritoneal Dialysis Patients
Brief Title: The Effect of Exercise on Blood Pressure Variability on Peritoneal Dialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Dong Sun, Clinical Professor, The Affiliated Hospital of Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: XWRCHT20210038
Record Dates: First submitted 2025-07-23; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D; Peritoneal Dialysis (PD)
Keywords: exercise; resistance; peritoneal dialysis; blood pressure; cardiovascular system; Blood Pressure Variability
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Exercise; Resistance Training

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Routine peritoneal dialysis care, health education, daily activity guidance, and dietary counseling were provided in accordance with the dietary guidelines for chronic kidney disease
- Exercise group (Experimental): Routine peritoneal dialysis care, health education, daily activity guidance, and dietary counseling were provided in a manner consistent with the care given to the control group-to avoid performance bias. In addition to routine basic care and treatment, the exercise group performed a combination of aerobic and resistance exercise
  Interventions: Behavioral: combination of aerobic and resistance exercise

INTERVENTIONS:
Behavioral: combination of aerobic and resistance exercise — Aerobic exercise: The main form is walking(gait), which includes three parts: warm-up, walking, and relaxation. Exercise time and frequency: 30-60 minutes of exercise per day, 3-5 times per week.
  Resistance exercise: Mainly uses elastic bands to enhance resistance exercise, since the risks of increased intra-abdominal pressure and fluid leakage in peritoneal dialysis patients is high, Investigator considered selective resistance exercise especially for limb and shoulder joint exercises. Patients can choose 3-5 muscle groups based on individual conditions, with each action 10-15 times and maintained for 10 seconds. Start with 2 sets of resistance exercise and then gradually increase to 3-5 sets, with 2-3 minutes of rest between each sets. Exercise frequency and duration: 2 times a week (non-consecutive days), 20 minutes each time.
  Other Names: Aerobic exercise; resistance exercise
  Arms: Exercise group

SUMMARY:
In China, the chronic kidney disease (CKD) incidence rate is as high as 10.8%. Renal replacement therapy plays an critical role in the later stage of CKD and becomes mandatory, as end-stage renal disease (ESRD) is unavoidable in progressive CKD. Peritoneal dialysis (PD) has becoming an essential alternative treatment for patient with end-stage renal disease (ESRD). Hypertension is common among ESRD patients receiving PD treatment, with a prevalence rate of 80% -90%, It is major cause for cardiovascular related complications and deaths among ESRD patients. Therefore hypertension increases the cardiovascular disease risk among the patients of ESRD and at the same time plays an independent risk for the progression of ESRD. Most studies uses average blood pressure as a risk indicator, but in recent years, more evidence has shown that blood pressure variability (BPV), the degree of fluctuation of blood pressure for a long period, is an additional risk factors for cardiovascular events.

DETAILED DESCRIPTION:
Cardiovascular events can be well predicted by Blood pressure variability (BPV) and is positively correlated with cardiovascular mortality, making it more informative than average blood pressure. BPV is also an excellent predictor of renal dysfunction and is significantly linked with the advancing renal insufficiency in CKD patients. Therefore, reducing BPV has important clinical significance for PD patients. At present, the research studies on impact of BPV in PD patients is very much limited, especially on the exercise impact on BPV in PD patients. Generally speaking the average physical activity in PD patients are well decreased. Low amount of exercise is correlated to high incidence rate and mortality of cardiovascular complication, depression, muscle atrophy, and eventually decreased quality of life. Relevant guidelines recommend that PD patients should engage in appropriate physical exercise to improve the outcome. Therefore, the purpose of this study is to investigate the effect of 12 week combined aerobic and resistance exercise on BPV in PD patients, in order to provide reference point for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis time ≥ 3 months, a stable condition;
* Age ≥ 18 years old;
* Hypertension (blood pressure>140 and/or 90 mmHg or currently under antihypertensive drugs), antihypertensive drugs was not changed or replaced during the complete trial;
* Patients with regular and sufficient peritoneal dialysis with kt/v>1.7, high compliance, and voluntary participation.

Exclusion Criteria:

* Blood pressure more than - systolic blood pressure ≥ 180mmHg, diastolic blood pressure ≥ 110mmHg;
* Severe anaemia Hb ≤ 60g;
* Cardiac function Class IV - In accordance with The New York Heart Association classification system, patients with severe cardiac disease resulting in inability to perform any physical activity without discomfort (If any physical activity is undertaken, discomfort is increased) or symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest.
* Using erythropoietin;
* There have been recent acute cardiovascular and cerebrovascular events, including vascular embolism, surgery, trauma, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
Difference between the coefficient of variation of mean daytime Systolic Blood Pressure from the baseline to the end of the study | Baseline/12Weeks
  Change in the coefficient of variation of mean daytime Systolic Blood Pressure as assessed by Ambulatory Blood Pressure Monitoring.
Difference between the Coefficient of variation of mean daytime Diastolic Blood Pressure from the baseline to the end of the study | Baseline/12Weeks
  Change in the Coefficient of variation of mean daytime Diastolic Blood Pressure as assessed by Ambulatory Blood Pressure Monitoring
Difference between the Coefficient of Variation of mean nighttime Systolic Blood Pressure from the baseline to the end of the study | Baseline/12Weeks
  Change in the Coefficient of Variation of mean nighttime Systolic Blood Pressure as assessed by Ambulatory Blood Pressure Monitoring
Difference between the Coefficient of Variation of mean nighttime Diastolic Blood Pressure from the baseline to the end of the study | Baseline/12Weeks
  Change in the Coefficient of Variation of mean nighttime Diastolic Blood Pressure as assessed by Ambulatory Blood Pressure Monitoring.

SECONDARY OUTCOMES:
Difference between the Coefficient of Variation of 24 Hours Systolic Blood Pressure from the baseline to the end of the study | Baseline/12Weeks
  Change in the Coefficient of Variation of 24 Hours Systolic Blood Pressure as assessed by Ambulatory Blood Pressure Monitoring.
Difference between the Coefficient of Variation of 24 Hours Diastolic Blood Pressure from the baseline to the end of the study | Baseline/12Weeks
  Change in the Coefficient of Variation of 24 Hours Diastolic Blood Pressure as assessed by Ambulatory Blood Pressure Monitoring.

CONTACTS AND LOCATIONS:
Locations (1):
- The affiliated hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China